CLINICAL TRIAL: NCT02623777
Title: Evaluation of the Effect of Arabinoxylan Oligosaccharides Consumption on Insulin Resistance in Patients With Metabolic Syndrome and the Contribution of Short-chain Fatty Acids Production
Brief Title: Effect of Arabinoxylan Oligosaccharides Consumption on Insulin Resistance in Patients With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kristin Verbeke, Prof. Kristin Verbeke, KU Leuven
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: s57413
Record Dates: First submitted 2015-11-28; First posted 2015-12-08 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Fatty Acids, Volatile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- AXOS as first intervention (Experimental): AXOS as first intervention
  Interventions: Dietary Supplement: Arabinoxylan oligosaccharides; Dietary Supplement: Short chain fatty acids
- SCFA as first intervention (Experimental): SCFA as first intervention
  Interventions: Dietary Supplement: Arabinoxylan oligosaccharides; Dietary Supplement: Short chain fatty acids

INTERVENTIONS:
Dietary Supplement: Arabinoxylan oligosaccharides — Arabinoxylan oligosaccharides administered
  Other Names: AXOS
Dietary Supplement: Short chain fatty acids — Short chain fatty acids administered
  Other Names: SCFA

SUMMARY:
During this project the investigators will evaluate whether the effects of arabinoxylan oligosaccharides (AXOS) consumption on insulin resistance in participants with metabolic syndrome can be explained by the production of short-chain fatty acids (SCFA). Secondly, the investigators will evaluate whether changes in gut hormone production might explain the effect on insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Regular diet (3 meals/day on at least 5 days/week)
* Central obese (defined as waist circumference ≥ 94cm for Europid men and ≥ 80cm for Europid women, with ethnicity specific values for other groups)
* Insulin resistant: HOMA-IR > 1.7 or fasting glucose > 100mg/dL
* And one of the following three factors:

  * Elevated TG level: ≥ 150 mg/dL (1.7 mmol/L)
  * Decreased HDL cholesterol level: < 40 mg/dL (1.03 mmol/L*) in males and < 50 mg/dL (1.29 mmol/L*) in females
  * Elevated blood pressure (BP): systolic BP ≥ 130 or diastolic BP ≥ 85 mm Hg

Exclusion Criteria:

* Low calorie diet or other special diet during the study or during the last month prior to the study
* Serious chronic disease of the gastrointestinal tract, such as inflammatory bowel disease (Crohn's disease or ulcerative colitis), irritable bowel syndrome, chronic constipation (less than 3 bowel movements a week), chronic frequent diarrhoea (more than 3 stools a day), clinically relevant lactose intolerance, …
* Use of antibiotics during the last month before starting the study
* Abdominal surgery in the past (except from appendectomy)
* Use of medication that affects the gastro-intestinal tract during the last 2 weeks prior to the study including spasmolytics, anti-diarrhoea medication, anti-constipation medication, and/or pre- or probiotic supplements (e.g. lacteol, Enterol)
* Pregnancy, pregnancy desire or lactation
* Diabetes (type 1 or 2), i.e. HbA1c > 6.5 %
* Abnormal haemoglobin (Hb) levels in blood, men must have an Hb level between 14.0 and 18.0 g / dL and women between 12.0 and 16.0 g / dL.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in insulin resistance after both interventions using the homeostatic model assessment for insulin resistance | 2 weeks